CLINICAL TRIAL: NCT03583788
Title: Effect of Hypnotherapy in Alcohol Use Disorder Compared to Motivational Interviewing. A Randomised Controlled Trial
Brief Title: Effect of Hypnotherapy in Alcohol Use Disorder Compared to Motivational Interviewing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HypnotherapyAUD
Record Dates: First submitted 2018-05-29; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Hypnosis; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: This study was designed as a parallel study, where two groups were compared: one receiving treatment as usual (motivational interviewing) and the intervention (hypnotherapy group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnotherapy group (Experimental): The intervention consisted of individual hypnotherapy of 5 hourly sessions (60 minutes) over 5 weeks, a total of five hours. The hypnotherapy treatment method was Erickson's (permissive) hypnosis (17). It began with a conversation about patient's past life events, present situation, alcohol problem and his or her thoughts about it. The hypnotherapy Group did not receive any treatment of motivational interviewing.
  Interventions: Behavioral: Hypnotherapy
- Motivational interviewing group (Active Comparator): The comparator patient group received individual therapy as motivational interviewing (MI) for 5 hourly sessions over 5 weeks, a total of five hours. The patients in the experimental group did not receive this.
  Interventions: Other: Motivational Interviewing

INTERVENTIONS:
Behavioral: Hypnotherapy — The intervention consisted of hypnotherapy given as five one-hour sessions over 5 weeks as individual therapy instead of motivational interviewing.
  Other Names: Motivational interviewing
  Arms: Hypnotherapy group
Other: Motivational Interviewing — The intervention consisted of Motivational Interviewing given as five one-hour sessions over 5 weeks as individual therapy instead of hypnotherapy.
  Arms: Motivational interviewing group

SUMMARY:
This study was carried out at an inpatient clinic in Norway. A six- week long treatment programme included intensive group therapy, but also five hours of individual therapy, given as motivational interviewing (MI). Thirty-one patients were randomized either to receive five individual sessions of hypnotherapy instead of MI (N=16) or to be in the control group (N=15). The treatment method for the hypnotherapy group was Erickson's (permissive) hypnosis. At baseline all the participants were diagnosed using a psychiatric interview and filled in the Alcohol Use Identification Test (AUDIT), Time-line-follow-back (TLFB) for alcohol use, Hopkins Symptoms Check List (HSCL-25) for monitoring mental distress and Traumatic Life Events Questionnaire. AUDIT, TLFB and HSCL-25 were re-administered at follow-up after one year.

DETAILED DESCRIPTION:
This study was designed as a parallel study, where two groups were compared: one receiving treatment as usual (motivational interviewing) and the intervention (hypnotherapy group). With difference in treatment effect as great as 40% we would have needed 46 participants to achieve p=0.05. We had initially planned to recruit as many as 50 individuals, but many were sceptical to the novel treatment. Four persons withdrew from the hypnotherapy group either before or after first treatment because of uncertainty. This did not affect randomization and they are not represented in the results.

Participants in the study were recruited from patients admitted to a six week long inpatient treatment programme at Vangseter Clinic in Norway in 2016. Only individuals who suffered from AUD were included in this study. The treatment programme consisted of the following elements: 5 hours of group therapy 5 days a week, a 2-3 day long family visit, where a family therapy session was also included, some obligatory group activities, like trips to museums or walks in nature, and lastly, informal activities, such as barbecues, watching movies together or discussions in the hall. All this was thought to contribute to the therapy of the patients. From the second week of the program the patients were expected to have one hour of additional individual therapy a week. It was conducted as motivational interviewing (MI), totaling five hours. MI is one of the most popular and effective modern treatments. As a brief intervention, MI appears to be at least as effective as, and possibly more effective than, other treatment methods. As an alternative to the MI sessions the patients enrolled in the study could receive five individual hour-long sessions of hypnotherapy.

Patients were informed about the study, were given time to consider, and if they volunteered to participate then signed a consent form. Thirty-one individuals, who took part in this randomized controlled trial (RCT), were assigned at random to receive either hypnotherapy (N=16) or to be in the control group (N=15).

At the beginning of the second week of treatment (baseline) all the participants were administered Mini International Neuro-psychiatric Interview (MINI) psychiatric interview to be able to diagnose mental problems other than AUD. Exclusion criteria were having psychotic episodes, a recent severe other psychiatric diagnosis or recent drug abuse other than alcohol.

In addition, all patients filled in the Alcohol Use Identification Test (AUDIT) and a Time-line-follow-back (TLFB) for registration of number of standardized alcohol units consumed and alcohol-related problems during the previous month. They also filled in the Hopkins Symptoms Check List (HSCL-25) to measure their level of mental distress. Mental distress was given as a global average of the HSCL-25 denoted Global Severity Index (GSI). The Traumatic Life Events Questionnaire was used to register traumatic life experiences. AUDIT, TLFB and HSCL-25 were re-administered one year later as a follow-up.

The intervention consisted of hypnotherapy given as five one-hour sessions over 5 weeks as individual therapy instead of motivational interviewing. The treatment method was Erickson's (permissive) hypnosis. Each treatment session began with a conversation about the patient's past life events, present situation, alcohol problem and his or her thoughts about it. To be able to use visualisation, patients were always asked when and where they bought alcohol, and how it was consumed. During the first part of the treatment session the theme of the hypnotic intervention was formulated, and then hypnotic trance was induced. The induction method was mostly a combination of relaxation and breathing exercises with mental pictures of a peaceful place. Once the trance was induced, the patient was asked to visualize mastery of a selected situation. This situation was tailored according to the patient's needs. It could include, for example, abstaining from alcohol at a party, passing an alcohol shop without going inside, or mastering another problematic issue, such as staying relaxed and calm in the presence of other people. When indicated, the events of the past were a subject of hypnotic intervention as well.

Data were analysed using Statistical Package for the Social Sciences (SPSS; IBM statistics) version 25, using simple bivariate analysis (Student's T-test or chi-square test), comparing the intervention group and the control group. Level of significance was set to p < 0.05, but even higher values were considered as the risk of type II statistical errors would be substantial in the small randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Only individuals who suffered from AUD were included in this study.

Exclusion Criteria:

* Exclusion criteria were having psychotic episodes, a recent severe other psychiatric diagnosis or recent drug abuse other than alcohol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Reduction of alcohol consumption | baseline + 12 months
  Alcohol consumption was measured at the entry to the study and at follow-up one year later using Alcohol Use Identification Test (AUDIT) registration of number of standardized alcohol units consumed and alcohol-related problems during the previous month.

SECONDARY OUTCOMES:
Level of mental distress | baseline + 12 months
  Mental distress was given as a global average of the HSCL-25 denoted Global Severity Index (GSI). HSCL-25 was administered at the entry to the study and at follow-up one year later

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen G Bramness, Ph.D., Study Director — Hospital Innlandet/ University of Tromso

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edwards G. Hypnosis in treatment of alcohol addiction. Controlled trial, with analysis of factors affecting outcome. Q J Stud Alcohol. 1966 Jun;27(2):221-41. No abstract available. PMID 5963138
- [Background] Hartman BJ. Hypnotherapeutic approaches to the treatment of alcoholism. J Natl Med Assoc. 1976 Mar;68(2):101-3, 147. No abstract available. PMID 1263266
- [Background] Pekala RJ, Maurer R, Kumar VK, Elliott NC, Masten E, Moon E, Salinger M. Self-hypnosis relapse prevention training with chronic drug/alcohol users: effects on self-esteem, affect, and relapse. Am J Clin Hypn. 2004 Apr;46(4):281-97. doi: 10.1080/00029157.2004.10403613. PMID 15190730
- [Background] Kohler S, Hofmann A. Can motivational interviewing in emergency care reduce alcohol consumption in young people? A systematic review and meta-analysis. Alcohol Alcohol. 2015 Mar;50(2):107-17. doi: 10.1093/alcalc/agu098. Epub 2015 Jan 6. PMID 25563299
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538